CLINICAL TRIAL: NCT02888496
Title: Caractérisation Des Anomalies Immunologiques au Cours de la Pseudopolyarthrite rhizomélique et Effets du Traitement Par Tocilizumab
Brief Title: Lymphocyte and Cytokine Disturbances in Polymyalgia Rheumatica
Acronym: TENOR-IMMUNO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TENOR-IMMUNO
Record Dates: First submitted 2016-08-26; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PMR patients: Patients included in the clinical trial TENOR (prospective open-labeled study of tocilizumab in treatment-naïve PMR patients)
  Interventions: Drug: tocilizumab
- Healthy controls: Matched to PMR patients for sex and age, exclusion of any autoimmune, inflammatory, neoplastic and chronic infectious disease

INTERVENTIONS:
Drug: tocilizumab — 3 monthly IV infusions in PMR patients
  Other Names: anti-IL-6 receptor monoclonal antibody
  Groups: PMR patients

SUMMARY:
Pathophysiology of polymyalgia rheumatica (PMR) is ill defined. This study aims at characterizing immunological abnormalities in PMR patients, and to assess the effects of tocilizumab therapy on this abnormalities.

DETAILED DESCRIPTION:
Comparison of PMR patients and matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

* PMR patient included in the TENOR study with samples available

Exclusion Criteria:

* Patient not included in the TENOR study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PMR patients included in the TENOR study (NCT01713842).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of blood lymphocyte populations (T cells, B cells, NK cells) | 6 months
  Lymphocyte subset analysis by flow cytometry

SECONDARY OUTCOMES:
Serum cytokine concentration measurement | 6 months
  Cytokine level measurements using an array and ELISAs

CONTACTS AND LOCATIONS:
Overall Officials: Divi Cornec, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devauchelle-Pensec V, Berthelot JM, Cornec D, Renaudineau Y, Marhadour T, Jousse-Joulin S, Querellou S, Garrigues F, De Bandt M, Gouillou M, Saraux A. Efficacy of first-line tocilizumab therapy in early polymyalgia rheumatica: a prospective longitudinal study. Ann Rheum Dis. 2016 Aug;75(8):1506-10. doi: 10.1136/annrheumdis-2015-208742. Epub 2016 Feb 29. PMID 26929219